CLINICAL TRIAL: NCT04371913
Title: Personalized Second Chance Breast Conservation (PSCBC): A Two Center Prospective Phase II Clinical Study
Brief Title: Personalized Second Chance Breast Conservation (PSCBC): A Prospective Phase II Clinical Study
Acronym: Second Chance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-07020531
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Radiation Therapy - PBI (Other): Patients will be treated with the fractionation of 30 Gy in 5 fractions over 1-2 weeks, which is the accelerated partial breast irradiation (PBI) fractionation scheme of choice for RT naïve patients at New York Presbyterian using External Beam Radiation Therapy (EBRT)
  Interventions: Radiation: 600cGY x 5 fractions APBI
- Radiation Therapy - WBRT (Other): Patients will be treated with the fractionation of 4050 cGy in 15 fractions over 3 weeks, which is the standard whole breast RT (WBRT) fractionation scheme of choice for RT naïve patients at New York Presbyterian using External Beam Radiation Therapy (EBRT)
  Interventions: Radiation: 270cGy x 15 fractions WBRT

INTERVENTIONS:
Radiation: 600cGY x 5 fractions APBI — Patients will be treated with the fractionation of 30 Gy in 5 fractions over 1-2 weeks, which is the accelerated fractionation scheme of choice for RT naïve patients at New York Presbyterian using EBRT
  Arms: Radiation Therapy - PBI
Radiation: 270cGy x 15 fractions WBRT — Patients will be treated with the fractionation of 4050 cGy in 15 fractions over 3 weeks, which is the standard whole breast RT (WBRT) fractionation scheme of choice for RT naïve patients at New York Presbyterian using External Beam Radiation Therapy (EBRT)
  Arms: Radiation Therapy - WBRT

SUMMARY:
The goal of the study is to investigate the feasibility of enabling a second chance for breast conservation in patients with in-breast recurrences after a previous lumpectomy and RT, investigators propose to test partial breast irradiation with the target volume encompassing the entire surgical bed with 1.0-1.5 cm margins.

An additional goal of the study is to investigate the feasibility of enabling a second chance for breast conservation in patients with inbreast recurrences after a previous lumpectomy and PBI, the investigators propose to test whole breast RT (WBRT) with the target as the whole breast volume.

DETAILED DESCRIPTION:
Patients will be treated with the fractionation of 30 Gy in 5 fractions over 1-2 weeks, which is the accelerated fractionation scheme of choice for Radiation Therapy (RT) naïve patients at New York Presbyterian using EBRT or with the fractionation of 4050 cGy in 15 fractions over 3 weeks, based on the previous treatment that they received.

The main aim of the study is to evaluate the rate of early grade 3 toxicities with this approach.

ELIGIBILITY:
Inclusion Criteria:

* Isolated ipsilateral unifocal breast lesions
* Limited size (< 2-3 cm) without evidence of skin involvement
* Histologically proven invasive breast carcinoma or carcinoma in situ
* Negative histologic margins of resection
* Patients with 0 to 3 positive axillary lymph nodes without extracapsular extension
* No synchronous distant metastases
* Age ≥ 18 years
* ≥ 12 months interval between initial breast conserving therapy (surgery and whole breast radiotherapy) and recurrence
* Previous WBI or IORT, brachytherapy or external beam partial breast treatment
* Technical feasibility
* Every kind of systemic therapy is allowed
* Informed consent for clinical and research purposes signed

Exclusion Criteria:

* Regional recurrences (axillary, supraclavicular)
* Positive histologic margins at resection
* Metastatic disease
* Poor cosmesis from previous surgery and RT
* Extensive Intraductal Component

Ages: 19 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment related adverse events as graded by CTCAE version 5.0 | up to 1 year from completion of radiation treatment
  The primary endpoint of the study is to test the feasibility in terms of acute toxicity of a protocol of partial breast re-irradiation for breast cancer treatment in a previously irradiated whole breast, as defined by the rate of grade ≥ 3 treatment-related skin, fibrosis, and breast pain AEs, as graded by CTCAE version 5.0.

SECONDARY OUTCOMES:
Number of participants with late toxicity will be measured as graded by CTCAE version 5.0 | up to 60 months
  Late toxicity is defined as the adverse events experienced by patients after 90 days post radiation therapy.
Change in number of participants with skin changes | baseline, approx. week 1- week 2 of radiation, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months.
  This count of participants will include patients who experience the following: skin hyperpigmentation, fibrosis, telangiectasia, skin induration and edema.
Change in Quality of life as assessed by Breast Cancer treatment outcome scale (BCTOS) | baseline, approx. week 1- week 2 of radiation, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months.
  The Breast Cancer Treatment Outcomes Scale (BCTOS) will be used to evaluate patient-reported cosmetic outcome, functional status, and breast pain. Each BCTOS subscale (cosmetic, functional status, and breast pain) is calculated by computing the arithmetic mean of the answers to each item relevant to a given subscale. The score is a continuous variable ranging from 1 to 4, with 1 indicating no difference between the treated and untreated breast, 2 indicating a slight difference, 3 indicating a moderate difference, and 4 indicating a large difference. Participants completing the BCTOS is optional.
Number of participants who demonstrate local control | 60 months
  Patients will be followed for recurrence of cancer in the treated breast.
Disease free survival (DFS) will be measured | 60 months
Overall Survival (OS) will be measured. | 60 months
Number of participants who received subsequent mastectomy in the treated breast | 6 months
  The investigators will track for enrolled patients the rate of subsequent mastectomy in the treated breast
Number of participants who received subsequent mastectomy in the treated breast | 12 months
  The investigators will track for enrolled patients the rate of subsequent mastectomy in the treated breast.
Number of participants who received subsequent mastectomy in the treated breast | 24 months
  The investigators will track for enrolled patients the rate of subsequent mastectomy in the treated breast.
Number of participants who received subsequent mastectomy in the treated breast | 36 months
  The investigators will track for enrolled patients the rate of subsequent mastectomy in the treated breast.
Number of participants who received subsequent mastectomy in the treated breast | 48 months
  The investigators will track for enrolled patients the rate of subsequent mastectomy in the treated breast.
Number of participants who received subsequent mastectomy in the treated breast | 60 months
  The investigators will track for enrolled patients the rate of subsequent mastectomy in the treated breast.

CONTACTS AND LOCATIONS:
Overall Officials: John Ng, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - New York Presbyterian Hospital - Queens, New York, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No